CLINICAL TRIAL: NCT01969318
Title: A Multicenter Randomized, Double-blind, Placebo Controlled ,Parallel Group ,Phase II Study to Access the Efficacy and Safety of SP2086 in Combination Therapy With Metformin in Patients With Type 2 Diabetes Patients
Brief Title: Efficacy and Safety Study of SP2086 in Combination With Metformin in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2086-202
Record Dates: First submitted 2013-10-17; First posted 2013-10-25 (Estimated); Last update posted 2013-10-25 (Estimated); Status verified 2013-10

CONDITIONS: Type 2 Diabetes
Keywords: SP2086; Phase II; combination therapy
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo/Metformin (Placebo Comparator)
  Interventions: Drug: Placebo /Metformin
- SP2086 (50mg q.d)/Metformin (Experimental)
  Interventions: Drug: SP2086(50 mg q.d.)/Metformin
- SP2086 (100mg q.d.)/Metformin (Experimental)
  Interventions: Drug: SP2086 (100 mg q.d.)/Metformin

INTERVENTIONS:
Drug: Placebo /Metformin — Patients are administered oral tablets of placebo once daily and metformin 500 mg t.i.d for 2 weeks at run-in period.After randomized,patients will be administered the drugs too
  Arms: Placebo/Metformin
Drug: SP2086(50 mg q.d.)/Metformin — patients are administered oral placebo once daily and metformin 500 mg t.i.d for 2 weeks at the run-in period .After randomized ,patients will be administered SP2086 50 mg q.d. and 500 mg t.i.d for 12 weeks
  Arms: SP2086 (50mg q.d)/Metformin
Drug: SP2086 (100 mg q.d.)/Metformin — patients are administered oral placebo once daily and metformin 500 mg t.i.d for 2 weeks at the run-in period .After randomized ,patients will be administered SP2086 100 mg q.d. and 500 mg t.i.d for 12 weeks
  Arms: SP2086 (100mg q.d.)/Metformin

SUMMARY:
SP2086 is a new dipeptidyl peptidase(DPP)-4 inhibitor. This study aims to evaluate the efficacy and safety of SP2086 in combination therapy with Metformin in patients with Type 2 Diabetes in Metformin monotherapy Who have Inadequate Glycemic Control

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with type 2 diabetes mellitus
* subject on metformin nontherapy with dose 1500mg/d for ≥12 weeks
* HbA1C：≥7.5% and ≤11.0%
* BMI:≥20 and ≤35 kg/m2

Exclusion Criteria:

1. <80% or >120% compliance with placebo treatment during the run-in period
2. Patients used the following drugs or therapies prior to randomization:

1) Somatropin therapy within 6 months prior to randomization 2) History of drug or alcohol abuse within 6 months prior to randomization 3) Participate in clinical trials of any drugs or medical devices within 3 months prior to randomization 4) Receive corticosteroids long-term (more than 7 consecutive days) oral, non-gastrointestinal administration or intra-articular administration within 2 months prior to randomization 5) Weight control drugs administration or Surgeries resulting in weight instability within 2 months prior to randomization 6) In investigator's opinion, patients used any drugs that interfere with assessment of the investigational product, or produce vital organs toxicity 4. Patients with history of the following diseases or proof prior to randomization:

1. Type 1 diabetes, single gene mutation diabetes, diabetes caused by pancreatic damage and secondary diabetes, such as caused by Cushing's syndrome or acromegaly
2. a history of hypertension, and after antihypertensive treatment, systolic blood pressure ≥ 160 mmHg or diastolic blood pressure ≥ 100 mmHg
3. a history of acute and chronic pancreatitis or pancreatic injury that may lead to high risk of pancreatitis
4. serious haematological diseases or other diseases leading to hemolyze and Red Blood Cell unstable (malaria、haemolytic anaemia eg. )
5. other endocrine diseases, for example hyperthyroidism、hypothyroidism、hypercortisolism、multiple endocrine neoplasia and so on
6. Any organ system tumors except the local skin basal cell carcinoma that have been treated or not been treated within 5 years prior to randomization, regardless of whether there is evidence of local recurrence or metastasis ; a history or family history of medullary carcinoma of thyroid ; a history of multiple endocrine neoplasia
7. Decompensated heart failure (NYHA class III and IV), unstable angina, stroke or transient ischemic attack, myocardial infarction, persistence and clinical significance arrhythmia, coronary artery bypass grafting or percutaneous coronary intervention within 6 months prior to randomization
8. Acute metabolic complications (ketoacidosis, lactic acidosis or hyperosmolar coma), unstable proliferative retinopathy or macular degeneration within 6 months prior to randomization
9. Severe trauma or acute infection that may affect blood glucose control within 4 weeks prior to randomization
10. Severe chronic gastrointestinal disease or therapy that may affect drug absorption, such as gastrointestinal surgery
11. With a history of mental/emotional disorder that would interfere with the subject's participation in the study.

5. Patients with any laboratory parameters meet the following criteria prior to randomization:

1. Aspartate Aminotransferase or alanine aminotransferase ≥ 2.0× upper normal limit(UNL) , and/or total bilirubin ≥ 2.0 × UNL also review confirmed within 3 days;
2. Triglyceride>5.64mmol/L（500mg/dl）；
3. serum creatinine to exceed the normal range
4. thyroid stimulating hormone to exceed the normal range, and have clinical significance
5. blood amylase o exceed the normal range, and have clinical significance
6. In investigator's opinion, any significant laboratory abnormalities of clinical significance value that interfere with assessment of this study.

6. At Screening patients not installed pacemaker with II or III degree atrioventricular block, long QT syndrome or QT corrected > 500 ms 7. Patients who received blood transfusions or blood donation≥ 400 mL or severe blood loss at least 400 mL within 8 weeks prior to randomization

-

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2012-03; Primary Completion 2012-08 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in HbA1c (Hemoglobin A1C) at Week 12 | baseline, week 12

SECONDARY OUTCOMES:
Percentage of Participants Achieving Less Than (<) 6.5% or <7% HbA1c Levels | week 12
Change From Baseline in Fasting Plasma Glucose at Week 4, 8 and 12 | Baseline, Week 4, 8, 12
Post-meal total and incremental glucose,insulin and C-peptide area under the curve at week 12 | baseline, week 12
Change from baseline in Homeostasis model assessment-beta(HOMA-β) at week12 | baseline, week 12
Change From Baseline in lipid at Week 12 | baseline, week12
Change From Baseline in Body Weight at Week 4,8,12 | baseline, Week 4, 8,12

CONTACTS AND LOCATIONS:
Overall Officials: Changyu Pan, M.D., Principal Investigator — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, China